CLINICAL TRIAL: NCT01905865
Title: The Role of Uncertainty in Coping Efficacy: The Experience of Parents of Children With Undiagnosed Medical Conditions
Brief Title: The Role of Uncertainty in Coping: The Experience of Parents of Children With Undiagnosed Medical Conditions
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Collaborators: University of Virginia (Other)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999913162; 13-HG-N162
Record Dates: First submitted 2013-07-18; First posted 2013-07-23 (Estimated); Last update posted 2026-01-28 (Actual); Status verified 2025-07-02

CONDITIONS: Undiagnosed Disease
Keywords: Undiagnosed Medical Conditions; Natural History
MeSH Terms: conditions — Undiagnosed Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parent: Persons aged 18 years or older who have a child with an undiagnosed medical condition, who have applied to the Undiagnosed Diseases Network, and have been assigned to the NIH.

SUMMARY:
Background:

- Parents of a child with an undiagnosed medical condition face a lot of uncertainty. They may not know how to take care of their child or how the illness will affect their family life. Researchers want to study how these parents cope with and adapt to their child s condition in light of this uncertainty. Being uncertain can make it hard for parents to adapt. But it also might give them hope. Researchers want to study how uncertain the parents think their situation is and how that affects the way they think they can cope. Personality traits, like being able to handle uncertainty and being resilient, might also affect coping.

Objectives:

- To understand how having a child with an undiagnosed illness affects the way their parents think they can cope.

Eligibility:

- Adults with a child who has a medical condition that has not been diagnosed for at least 2 years and involves at least 2 parts of the body.

Design:

* Participants will answer survey questions for about 30 minutes. The questions are about their thoughts and feelings about having a child with an undisclosed illness.
* Participants can take the survey on paper or online.

DETAILED DESCRIPTION:
The proposed study aims to test the effect of the degree of perceived uncertainty on coping efficacy among parents of children with undiagnosed medical conditions. There are many dimensions to uncertainty when there is no identified cause for a condition that affects one s child. They include illness identity, management, longevity and life planning, the meaning of the child s condition for the family and both the child s and the family s social connections. How parents of children with undiagnosed medical conditions appraise, cope and ultimately adapt to their child s condition in light of this uncertainty is largely unexplored. While high levels of perceived uncertainty may be seen as a threat to adaptation, there is evidence that parents find hope and opportunity in the uncertainty. The literature suggests that many factors affect how uncertainty is appraised, and higher levels of coping self-efficacy are associated with more effective coping and ultimately better adaptation. There is no research that systematically assesses the dimensions of uncertainty perceived by parents and whether overall perceptions of uncertainty or particular subsets are associated with coping efficacy. Further, personality traits, such as tolerance of uncertainty and resilience, may moderate these unexplored relationships. This study s conceptual framework is based on Lazarus and Folkman s Transactional Model of Stress and Coping and Mishel s Perceived Uncertainty in Illness Theory. A cross-sectional survey design will be used to quantitatively assess the relationships between dimensions of uncertainty and coping efficacy. Participants will be recruited through online support groups, website postings, and listservs. They will have the option of completing either a paper or online version of the survey.

ELIGIBILITY:
* Participants for this study will be English speaking men and women ages 18 years or older who have a child with an undiagnosed medical condition who have applied to the Undiagnosed Diseases Network, and have been assigned to the NIH.

The participant may be the adoptive or biological parent.

Parents may decide between themselves who will complete the survey as only one survey per household will be allowed.

Ages: 18 Years to 115 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants for this study will be English speaking men and women ages 18 years or older who have a child with an undiagnosed medical condition, who have applied to the Undiagnosed Diseases Network, and have been assigned to the NIH.
Sampling Method: Non-Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2013-06-12; Primary Completion 2013-06-12 (Actual)

PRIMARY OUTCOMES:
A | Enrollment
  To assess the dimensions of perceived uncertainty and their relative importance among parents of children with undiagnosed medicalconditions.
B | Enrollment
  To assess the role of uncertainty in predicting coping efficacy among parents of children with undiagnosed medical conditions.
C | Enrollment
  To determine whether tolerance for uncertainty and optimism moderate the relationship between uncertainty and coping efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Ellen F Macnamara, Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Human Genome Research Institute (NHGRI), 9000 Rockville Pike, Bethesda, Maryland, United States